CLINICAL TRIAL: NCT05969756
Title: Clinical Effectiveness of Early Treatments for Preventing Occlusal Caries Lesions in Erupting Permanent Molars
Brief Title: Early Treatments for Preventing Occlusal Caries Lesions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hue University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Le Van Nhat Thang, DDS, PhD, Principal Investigator, Hue University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H2023/012
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Caries; Initial; Occlusal Caries; Caries,Dental
Keywords: early caries lesions; sealants; erupting molars
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: This is a 3 arm clinical trial. All selected permanent molars will be randomly equally allocated into three groups according to material used.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of examiners is impossible to be done during intervention and follow up due to different natures of the materials. However, participants and outcome assessors could be blinded (double blinding).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fluoride varnish group (Experimental): 5% sodium fluoride varnish, 3M, USA
  Interventions: Drug: Fluoride varnish
- Conventional etch and rinse sealant group (Experimental): Resin-based composite sealant, 3M, USA
  Interventions: Drug: Conventional etch and rinse sealant
- Self-etch sealant group (Active Comparator): Self-etch primed sealant, Shofu, Japan
  Interventions: Drug: Self-etch sealant

INTERVENTIONS:
Drug: Fluoride varnish — Thirty-eight permanent molars will receive 5% sodium fluoride varnish application every three months
  Other Names: 3M™ Clinpro™ White Varnish
  Arms: Fluoride varnish group
Drug: Conventional etch and rinse sealant — Thirty-eight permanent molars will receive conventional etch and rinse sealant
  Other Names: 3M™ Clinpro™ Sealant
  Arms: Conventional etch and rinse sealant group
Drug: Self-etch sealant — Thirty-eight permanent molars will receive self-etch sealant
  Other Names: S-PRG filler-containing resin sealant; Beautisealant
  Arms: Self-etch sealant group

SUMMARY:
Sealants effectively arrest non-cavitated caries lesions on the fully erupted occlusal surface of permanent teeth. However, the clinical effectiveness of sealants is uncertain in preventing occlusal caries lesions in partially erupted permanent molars. This study aims to evaluate the progression of caries, the degree of retention, survival rate, and quality of the remnant after applying conventional total-etch resinous sealant and self-etch sealant in erupting molars.

ELIGIBILITY:
Inclusion Criteria:

For children:

1. Children presenting with good general health and cooperative behavior.
2. Children having early caries lesions in a permanent molar (first or second).
3. Parents signed informed consent.

For permanent molars:

1. Early caries lesions on the occlusal surface corresponding to International Caries Detection and Assessment System (ICDAS) scores 1 and 2. [Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8].
2. Erupting molars: eruption stages 2 (fully erupted occlusal surface with less than half of the crown exposed) and 3 (fully erupted occlusal surface with more than half of the crown exposed). [Carvalho JC, Ekstrand KR, Thylstrup A. Dental plaque and caries on occlusal surfaces of first permanent molars in relation to stage of eruption. J Dent Res. 1989 May;68(5):773-9].

Exclusion Criteria:

For children:

1. Any allergy reported by the parents.
2. Children unable to return for recall visits.

For permanent molars:

1. Teeth with occlusal surfaces completely covered by the gingival tissue.
2. Teeth with hypoplastic defects, restorations, or sealants.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 114 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Development of new caries lesion | 3 months
  ICDAS was considered "0'' for fully sealed teeth. A score of ICDAS≥1 was considered as new caries lesion
Development of new caries lesion | 6 months
  ICDAS was considered "0'' for fully sealed teeth. A score of ICDAS≥1 was considered as new caries lesion
Development of new caries lesion | 9 months
  ICDAS was considered "0'' for fully sealed teeth. A score of ICDAS≥1 was considered as new caries lesion
Development of new caries lesion | 12 months
  ICDAS was considered "0'' for fully sealed teeth. A score of ICDAS≥1 was considered as new caries lesion

SECONDARY OUTCOMES:
Sealants retention | 3 months
  Sealant retention was assessed as follows: total retention of sealant on the occlusal surface or the partial or complete absence of the sealant on the occlusal surface.
Sealants retention | 6 months
  Sealant retention was assessed as follows: total retention of sealant on the occlusal surface or the partial or complete absence of the sealant on the occlusal surface.
Sealants retention | 9 months
  Sealant retention was assessed as follows: total retention of sealant on the occlusal surface or the partial or complete absence of the sealant on the occlusal surface.
Sealants retention | 12 months
  Sealant retention was assessed as follows: total retention of sealant on the occlusal surface or the partial or complete absence of the sealant on the occlusal surface.
Quality of sealants | 3 months
  Quality of the remnant United States Public Health Service criteria (USPHS): anatomical shape, marginal adaptation, surface texture, and marginal discoloration.
Quality of sealants | 6 months
  Quality of the remnant United States Public Health Service criteria (USPHS): anatomical shape, marginal adaptation, surface texture, and marginal discoloration.
Quality of sealants | 9 months
  Quality of the remnant United States Public Health Service criteria (USPHS): anatomical shape, marginal adaptation, surface texture, and marginal discoloration.
Quality of sealants | 12 months
  Quality of the remnant United States Public Health Service criteria (USPHS): anatomical shape, marginal adaptation, surface texture, and marginal discoloration.

CONTACTS AND LOCATIONS:
Overall Officials: Van Nhat Thang Le, DDS, PhD, Principal Investigator — Hue University of Medicine and Pharmacy
Locations (2):
- Vietnam (2):
  - Hue University of Medicine and Pharmacy, Huế, Thừa Thiên Huế Province
  - Phu Vang Hospital, Phú Vang, Thừa Thiên Huế Province

IPD SHARING:
Plan to Share IPD: Yes
Will plan to share information when finishing study
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Plan to complete study in 1 year and will share the data after get publication